CLINICAL TRIAL: NCT05126277
Title: A Randomized, Double-blind, Parallel Group, Placebo-controlled, Multicenter Phase 3 Trial to Evaluate Efficacy, Safety and Tolerability of Ianalumab on Top of Standard-of-care Therapy in Participants With Active Lupus Nephritis (SIRIUS-LN).
Brief Title: Safety, Efficacy and Tolerability of Ianalumab Versus Placebo, Combination With SoC Therapy, in Participants With Active Lupus Nephritis
Acronym: SIRIUS-LN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736K12301; 2020-005830-14 (EudraCT Number); 2023-508559-37-00 (Other: EU CTIS)
Record Dates: First submitted 2021-10-15; First posted 2021-11-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lupus Nephritis
Keywords: SLE; Systemic Lupus Erythematosus (SLE); Kidney inflammation; Anti-BAFF-receptor; B cell depletion; Ianalumab; VAY736
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic; Nephritis | interventions — ianalumab

STUDY DESIGN:
Intervention Model Description: This is a pivotal double-blind, randomized, placebo-controlled, multi-center three-arm study, evaluating at Week 72 efficacy and safety of ianalumab administered s.c. every 4 weeks or ianalumab administered s.c. every 12 weeks versus placebo, administered s.c. every 4 weeks, in adult participants with active LN receiving SoC. In addition, long-term efficacy, safety and tolerability will be collected up to Week 144.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 - ianalumab s.c. q4w (Experimental): ianalumab s.c. q4w in addition to standard of care (SoC)
  Interventions: Drug: ianalumab s.c. q4w
- Arm 2 - ianalumab s.c. q12w (Experimental): ianalumab s.c. q12w in addition to SoC
  Interventions: Drug: ianalumab s.c. q12w
- Arm 3 - placebo s.c. q4w (Placebo Comparator): Placebo s.c. q4w in addition to SoC
  Interventions: Drug: placebo s.c.

INTERVENTIONS:
Drug: ianalumab s.c. q4w — ianalumab s.c. q4w in addition to SoC
  Other Names: VAY736
  Arms: Arm 1 - ianalumab s.c. q4w
Drug: ianalumab s.c. q12w — ianalumab s.c. q12w in addition to SoC
  Other Names: VAY736
  Arms: Arm 2 - ianalumab s.c. q12w
Drug: placebo s.c. — placebo s.c. q4w in addition to SoC
  Other Names: placebo
  Arms: Arm 3 - placebo s.c. q4w

SUMMARY:
This trial will evaluate efficacy, safety, and tolerability of subcutaneous (s.c.) ianalumab given every 4 weeks (q4w) or every 12 weeks (q12w) compared to placebo, in combination with SoC, in adult participants with active LN

DETAILED DESCRIPTION:
This trial will evaluate the efficacy, safety, and tolerability of subcutaneous (s.c.) ianalumab given every 4 weeks (q4w) or ianalumab given every 12 weeks (q12w) compared to placebo, in combination with SoC, in adult participants with active LN (ISN/RPS class III, IV active glomerulonephritis with or without co-existing class V features, or pure class V membranous). using the 2003 International Society for Nephrology (ISN)/Renal Pathology Society (RPS) criteria).

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

* Adult male and female participants aged 18 years or older at the time of screening
* Weigh at least 35 kg at screening
* Have a confirmed clinical diagnosis of SLE according to European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) Systemic Lupus Erythematosus (SLE) classification criteria
* Have a positive anti-nuclear antibody (ANA) test result; ANA titer ≥ 1:80 at screening visit based on central or local laboratory result
* Active LN at screening, as defined by meeting the 3 following criteria:
* Renal biopsy within 6 months prior to screening period indicating ISN/RPS class III or IV active glomerulonephritis with or without co-existing class V features, or pure class V membranous LN. If no biopsy was performed within 6 months prior to screening period, a biopsy will need to be performed during the screening period after having met all other inclusion/exclusion criteria.
* UPCR ≥ 1.0 g/g on 24h urine collection at Screening
* eGFR ≥ 25mL/min/1.73 m2. Participants with eGFR < 30 mL/min/1.73 m2 require renal biopsy during the screening period showing sclerosis in ≤ 50% of glomeruli
* Newly diagnosed participants as well as pre-treated LN participants (including refractory cases) can be included, as long as they are currently on, or willing to initiate SoC induction therapy for LN using MPA

  * Induction therapy, as defined by treatment including both high dose corticosteroids and MPA, should be initiated prior to or on day of randomization
  * Anti-malarial treatment at stable dosing prior to randomization is strongly recommended, in the absence of contraindications
  * Participants on azathioprine treatment at Screening must be switched to MPA prior to randomization
* Receipt of at least one dose of pulse methylprednisolone i.v. (250 - 1000 mg per day up to 3000 mg cumulative dose) or equivalent for treatment of current episode of active LN within 60 days prior randomization. Participant who cannot take the pulse i.v. corticosteroid therapy should directly start on 0.8-1.0 mg/day (max 80mg/day) oral predniso(lo)ne.
* Able to communicate well with the Investigator to understand and comply with the requirements of the study

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study:

* Severe renal impairment as defined by i.) presence of oliguria (defined as a documented urine volume <400 mL/24 hrs) or ii.) End-Stage Renal Disease (ESRD) requiring dialysis or transplantation
* Sclerosis in > 50% of glomeruli on renal biopsy
* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days or until the expected pharmacodynamic effect has returned to baseline. Use of certain Traditional Chinese Medicines
* Prior use of ianalumab (ever); or prior use other B cell depleting therapy within 36 weeks prior to randomization or if therapy was administered < 36 weeks prior to randomization, B cell count less than the lower limit of normal or patient's own baseline value prior to having received an earlier B cell-depleting therapy
* Prior treatment with any of the following within 12 weeks prior to randomization

  * Belimumab, telitacicept, abatacept, TNF-α mAb, immunoglobulins (i.v./s.c.) plasmapheresis
  * Any other immuno-suppressants (i.v. or oral cyclophosphamide, calcineurin inhibitors, JAK inhibitors or other kinase inhibitors)
  * Thalidomide treatment and/or methotrexate
  * Combination of DMARDs
* Imidazole derivative (e.g., azathioprine, mizoribine) must be discontinued prior to starting treatment with MPA
* Receipt of more than 3000 mg i.v. pulse methylprednisolone (cumulative dose) within 12 weeks prior to randomization
* History of major organ transplant or hematopoietic stem cell/bone marrow transplant or are due to receive transplantation
* Any one of the following laboratory values at screening:

  * Hemoglobin levels < 8.0 g/dL (< 5 mmol/L), or < 7.0 g/dL (< 4.3 mmol/L) if related to participant's SLE such as in active hemolytic anaemia
  * Platelet count < 25 x 1000/µL
  * Absolute neutrophil count (ANC) < 0.8 x 1000/µL
* Active viral, bacterial or other infections requiring intravenous or intramuscular treatment for clinically significant infection or history of recurrent clinically significant infection which in the opinion of the investigator will place the participant at risk for participation.
* History of known intolerance/hypersensitivity to MPA, oral corticosteroids, or any component of the study drug(s) or its excipients
* Receipt of live/attenuated vaccine within a 4-week period prior to randomization
* History of primary or secondary immunodeficiency, including a positive HIV test result
* History of malignancy of any organ system (other than localized basal cell carcinoma or squamous cell carcinoma of the skin or or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
* Any surgical, medical (e.g., uncontrolled hypertension, heart failure or diabetes), psychiatric or additional physical condition that the Investigator feels may jeopardize the participants in case of participation in this study
* Chronic infection with hepatitis B (HBV) or hepatitis C (HCV). Positive serology for hepatitis B surface antigen (HBsAg) excludes the participant
* Evidence of active tuberculosis (TB) infection (after anti-TB treatment, participants with history of TB may become eligible according to national local guidelines)
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 6 months after stopping of investigational medication
* Sexually active male participants, who do not agree to use barrier protection during intercourse with women of child-bearing potential while taking study treatment

Other protocol -defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2027-06-22 (Estimated); Study Completion 2030-11-05 (Estimated)

PRIMARY OUTCOMES:
Frequency and percentage of participants achieving stable Complete Renal Response (CRR) | Week 72
  The primary objective is to demonstrate superiority of ianalumab compared to placebo, in achieving stable CRR (defined as estimated glomerular filtration rate (eGFR) ≥90 ml/min/1.73 m2 or no less than 85% of baseline, AND, 24-hour UPCR <0.5 g/g) at Week 72 in active lupus nephritis (ISN/RPS class III, IV active glomerulonephritis with or without co-existing class V features, or pure class V membranous) participants on background SoC therapy.

SECONDARY OUTCOMES:
Time to first occurrence of stable urine protein-to-creatinine ratio (UPCR) <0.5 g/g or ≥50% reduction from baseline | Week 72
  To demonstrate superiority of ianalumab, compared to placebo, in time to first occurrence of stable urine protein-to-creatinine ratio (UPCR) <0.5 g/g or ≥50% reduction from baseline up to Week 72
Percentage of participants achieving stable Overall Renal Response (ORR), defined as achievement as either Complete Renal Response (CRR) or Partial Renal Response (PRR) | Week 48
  To demonstrate superiority of ianalumab, compared to placebo, in achieving stable Overall Renal Response (ORR) at Week 48
Incidence of stable Complete Renal Response (CRR) while maintaining daily corticosteroid dose ≤5 mg/day | Week 72
  To demonstrate superiority of ianalumab, compared to placebo, in achieving stable Complete Renal Response (CRR) at Week 72 while maintaining daily corticosteroid dose ≤5 mg/day between Week 24 and Week 72
Incidence of renal-related event or death | Week 72
  To demonstrate superiority of ianalumab, compared to placebo, in preventing renal-related event or death through Week 72
Change in British Isles Lupus Activity Group (BILAG) score | Week 72
  To demonstrate superiority of ianalumab, compared to placebo in BILAG-2004 at Week 72
Change in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue score | Week 72
  To demonstrate superiority of ianalumab, compared to placebo, in FACIT-Fatigue at Week 72
Number of participants with treatment-emergent Adverse Events (AEs) | Week 72
  AEs are any untoward sign or symptom that occurs during the study treatment
Ianalumab concentration in serum | Week 72
  To characterize the pharmacokinetics (PK) of ianalumab mean, median, minimum and maximum concentrations will be provided
Incidence and titer of anti-ianalumab antibodies in serum (ADA assay) over time | Week 72
  To evaluate immunogenicity of ianalumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (164):
- United States (37):
  - University Of Alabama, Birmingham, Alabama
  - Advanced Medical Research, La Palma, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - University of California LA, Los Angeles, California
  - University of California Irvine, Orange, California
  - School Of Medicine, Sacramento, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University Of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Fides Clinical Research, Atlanta, Georgia
  - Parris and Associates Rheumatology, Lawrenceville, Georgia
  - University of Kansas Hospital, Kansas City, Kansas
  - Accurate Clinical Research, Lake Charles, Louisiana
  - UMC New Orleans, New Orleans, Louisiana
  - Wayne State University, Detroit, Michigan
  - Univ of Nevada School of Med, Las Vegas, Nevada
  - Sahni Rheumatology and Therapy, West Long Branch, New Jersey
  - VA NM Healthcare System, Albuquerque, New Mexico
  - NY Nephrology, Clifton Park, New York
  - Hospital for Special Surgery, New York, New York
  - Northwell Health, New York, New York
  - Circuit Clinical, Orchard Park, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Brookview Hills Research Assoc, Winston-Salem, North Carolina
  - University Of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Arthritis and Rheumatology Ins, Allen, Texas
  - Precision Comprehensive Research, Colleyville, Texas
  - Liberty Research Center, Dallas, Texas
  - Univof Texas Southwestern Med Cntr, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Uni of Texas Health Science Center, San Antonio, Texas
  - Baylor Scott and White Research, Temple, Texas
  - Northern Assoc of Northern VA, Fairfax, Virginia
  - Uni Wisconsin School Med Pub Health, Madison, Wisconsin
- Argentina (6):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, San Miguel de Tucumán
- Brazil (10):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, São Luís, Maranhão
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Salvador
- Canada (8):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Chile (2):
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Temuco
- China (21):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Liuchow, Guangxi
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Binzhou, Shandong
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Colombia (3):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogota, Cundinamarca
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Tallinn, Estonia
- France (9):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (4):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Münster
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City
  - Novartis Investigative Site, Quetzaltenango
- Hong Kong (2):
  - Novartis Investigative Site, Kwun Tong, Kowloon
  - Novartis Investigative Site, Tuenmen
- Hungary (3):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kaposvár
- India (4):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Secunderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Chandigarh
- Italy (9):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Napoli
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Sibu, Sarawak
  - Novartis Investigative Site, Kuala Terengganu, Terengganu
- Mexico (4):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Oaxaca City
  - Novartis Investigative Site, Querétaro
- Romania (5):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Oradea, Jud Bihor
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Râmnicu Vâlcea, Vâlcea County
  - Novartis Investigative Site, Bucharest
- Novartis Investigative Site, Singapore, Singapore
- South Korea (7):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Daejeon, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (9):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (2):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, London
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com